CLINICAL TRIAL: NCT07318987
Title: EFFECT OF SAPHENOUS NERVE RELEASE ON PAIN,BALANCE AND FUNCTION IN PATIENTS WITH PATELLOFEMORAL PAIN SYNDROME
Brief Title: EFFECT OF SAPHENOUS NERVE RELEASE ON PATIENTS WITH PATELLOFEMORAL PAIN SYNDROME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Markos Boshra Agaiby Amin, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006114
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: PATELLOFEMORAL PAIN SYNDROME; Balance; pain; knee function; saphenous nerve
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Saphenous nerve release
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAPHENOUS NERVE RELEASE (Experimental): The patient is in a supine position with the leg extended. Look for a sensitive area four to five fingerbreadths above the knee on the medial side. This will be a long strip of fascia that is several inches in length. The fingers are then placed on either side of this strip on the medial side of the leg behind the sartorius muscle. The fingers are pulled apart in distal and proximal directions, as if to separate the strip as far as possible
  Interventions: Other: Saphenous nerve release
- traditional treatment (Active Comparator): The intervention program lasted six weeks and was performed three times per week. It included strengthening, manual therapy, and stretching exercises. Strengthening focused on both the hip and knee. Hip exercises consisted of side-lying hip abduction, clamshells, and prone hip extension, while knee exercises included straight leg raises, terminal knee extensions, and wall-supported mini-squats. Exercises progressed from 3 sets of 10 to 3 sets of 20 repetitions, with gradual resistance added, dynamic execution, brief pauses between repetitions, and short rest periods between sets.
  Manual therapy involved patellofemoral joint mobilization performed in a supine position with the knee slightly flexed, using superior, inferior, medial, and lateral patellar glides.
  Stretching exercises were performed in sitting or standing, targeting the posterior structures with the knee extended and ankle dorsiflexed. Static stretches were held for 15 seconds and repeated for three sets.
  Interventions: Other: Saphenous nerve release

INTERVENTIONS:
Other: Saphenous nerve release — With the patient lying supine and the leg extended, a tender area is identified on the medial side of the thigh, approximately four to five fingerbreadths above the knee. This area corresponds to a longitudinal fascial strip located behind the sartorius muscle. The therapist places the fingers on either side of this strip and applies a gentle separating force in proximal and distal directions to mobilize the tissue and reduce sensitivity.

SUMMARY:
Patellofemoral Pain Syndrome (PFPS) is a frequent cause of anterior knee pain in young, physically active individuals, especially females, and is commonly managed with quadriceps and hip-focused exercises. However, the role of neural factors has been largely overlooked. The saphenous nerve, which supplies sensation to the anteromedial knee, may become irritated or entrapped and contribute to pain and neuromuscular dysfunction in PFPS. This study suggests that manual therapy targeting the saphenous nerve could improve pain, function, and balance, providing a more holistic approach to PFPS rehabilitation.

DETAILED DESCRIPTION:
Patellofemoral Pain Syndrome (PFPS) is a common cause of anterior knee pain, particularly affecting adolescents and young adults, with a higher prevalence among females. It accounts for a significant proportion of knee complaints seen in sports medicine and is especially common in physically active individuals. Traditional rehabilitation for PFPS has mainly focused on quadriceps strengthening and knee mechanics, with more recent attention given to hip-focused exercises.

However, the neural contribution to PFPS, particularly involving the saphenous nerve and its infrapatellar branch, has been relatively under-explored. The saphenous nerve is a purely sensory branch of the femoral nerve that supplies the anteromedial knee and lower leg and plays an important role in proprioception. Anatomical variations and its course near the sartorius muscle may predispose it to irritation or entrapment, potentially contributing to chronic anteromedial knee pain.

This study proposes that irritation or mechanosensitivity of the saphenous nerve may be a contributing factor in PFPS, leading to pain and impaired neuromuscular control. By incorporating manual therapy targeting the saphenous nerve, the research aims to fill a gap in current PFPS management. Addressing neural factors may enhance pain reduction, functional performance, and balance, offering a more comprehensive and holistic physiotherapy approach for individuals with PFPS. (summarize in short)

ELIGIBILITY:
Inclusion Criteria:

1 - Age from 18 to 35 and BMI 18 to 25 kg/m2. 2. Both gender (male and female) 3. Patients who had anterior knee pain for at least six weeks 4. Patients with positive saphenous neurodynamic test (SAPHNT)

Exclusion Criteria:

1. Knee replacement
2. An intraarticular injection within the past 3 months
3. Previous operative treatment or arthroscopy, other secondary knee-related problems (bursitis, tendinopathy, osteochondritis, neuromas, intraarticular pathology (such as osteoarthritis), tumor, and rheumatologic diseases
4. Diabetic neuropathic pain or fibromyalgia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
knee pain | up to 6 weeks
  Visual analogue scale to measure pain intensity
Balance | up to 6 weeks
  Using the Biodex Stability System (Biodex balance system), static balance was measured
Function | up to 6 weeks
  Kujala Anterior Knee Pain Scale (AKPS) for knee pain and function, The Kujala score is composed of 13 multiple choice questions: the presence of a limp, the need for support, the ability to walk, the ability to climb stairs, the ability to squat, the ability to run, the ability to jump, prolonged sitting with knees in the flexed position, the presence of knee pain, the presence of knee swelling, the presence of abnormal painful patellar movement, atrophy of the thigh muscles, and deficiency of knee flexion.

SECONDARY OUTCOMES:
Q angle | up to 6 weeks
  The Q-angle is the angle formed between a line from the anterior superior iliac spine (ASIS) to the center of the patella and a line from the center of the patella to the tibial tuberosity. It reflects the alignment of the quadriceps muscle and the patellofemoral joint and is commonly assessed in patients with PFPS.
  Kinovea can be used to measure the Q-angle accurately by placing visual markers on the ASIS, patellar center, and tibial tuberosity, then capturing a frontal-plane image or video. Using Kinovea's angle measurement tool, the two lines are drawn and the angle is calculated. This provides a valid, reliable, and non-invasive method for assessing Q-angle in clinical and research settings, particularly for evaluating lower-limb alignment in PFPS.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided